CLINICAL TRIAL: NCT03471663
Title: A Phase I, Open-Label Study of D-0502 Single Agent and D-0502 in Combination With Palbociclib in Women With Advanced or Metastatic ER-Positive and HER2-Negative Breast Cancer
Brief Title: A First-in-Human Study of D-0502 Alone and in Combination With Palbociclib in Women With Advanced or Metastatic ER-Positive and HER2-Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBIO-301
Record Dates: First submitted 2018-03-14; First posted 2018-03-20 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- D-0502 (Experimental): D-0502
  Interventions: Drug: D-0502
- D-0502 in combination with palbociclib (Experimental): D-0502 in combination with palbociclib
  Interventions: Drug: D-0502; Drug: palbociclib

INTERVENTIONS:
Drug: D-0502 — oral tablets
Drug: palbociclib — standard dose of palbociclib
  Arms: D-0502 in combination with palbociclib

SUMMARY:
This is a phase I, open-label study of D-0502 single agent and D-0502 in combination with standard dose of palbociclib to assess the safety and tolerability, identify an MTD, and/or RP2D, evaluate the PK properties and evaluate preliminary anti-tumor activities in women with advanced or metastatic ER-positive, HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-proven, ER-positive, HER2-negative locally advanced, inoperable, and/or metastatic breast cancer.
2. Female patients with menopausal status:

   i. Postmenopausal status defined as meeting at least one of the following criteria:
   1. Have undergone a bilateral oophorectomy any time in life;
   2. Age ≥60 years, or
   3. Age <60 years but have cessation of regular menses ≥12 months with follicle stimulating hormone (FSH) value >40 milli-international units per milliliter (mIU/mL) and an estradiol value <40 picograms per milliliter (pg/mL) (140 picomoles per liter [pmol/L]).

   ii. Premenopausal or perimenopausal concurrently given a luteinizing hormone-releasing hormone (LHRH) agonist starting at least 4 weeks before the start of trial therapy and is planned to continue LHRH agonist during the study.
3. Patients meeting all the following criteria:

   1. Has had at least 6 months of endocrine therapy for metastatic ER+ breast cancer prior to disease progression;
   2. Limited number of prior chemotherapy, endocrine therapy, and targeted therapy for advanced or metastatic disease
   3. Radiological or objective evidence of disease progression on or after the last systemic therapy prior to starting current study treatment.
   4. For phase Ia: Not eligible for standard therapy that would confer clinical benefit to the patient.

Exclusion Criteria:

1. Patients with prior anticancer or investigational drug treatment within the following windows are excluded:
2. Participants with prior anticancer or investigational drug treatment within the following windows are excluded:

   1. Any anti-cancer therapy (including endocrine therapy, chemotherapy, targeted therapy, etc.) less than 30 days before first dose of study treatment.
   2. Any investigational drug therapy less than 28 days or 4 half-lives (whichever is shorter) prior to first dose of study treatment.
3. Patients with untreated or symptomatic or progressive central nervous system (CNS) metastases.

   * Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-03-18 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs meeting protocol defined dose-limiting toxicities (DLTs) criteria | Approximately 2 years

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) | Cycle 1 (28 days)
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] | Cycle 1 (28 days)
Time of maximum observed concentration (Tmax) | Cycle 1 (28 days)
Objective response rate (ORR) | up to 12 months
Progression free survival (PFS) | up to 12 months

CONTACTS AND LOCATIONS:
Locations (14):
- United States (10):
  - Local Institution, Fresno, California
  - Local Institution, Aurora, Colorado
  - Local Institution, New Haven, Connecticut
  - Local Institution, Boston, Massachusetts
  - Local Institution, Eugene, Oregon
  - Local Institution, Greenville, South Carolina
  - Local Institution, Nashville, Tennessee
  - Local Institution, Dallas, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Tyler, Texas
- China (4):
  - Local Institution, Beijing, Chaoyang District
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Changsha, Hunan Provence
  - Local Institution, Shenyang, Liaoning